CLINICAL TRIAL: NCT00212355
Title: Phase3, Open-Label, Clinical Trial of Zinc Acetate for Treatment of Wilson's Disease in Japan.
Brief Title: Efficacy and Safety, Long-term Study of Zinc Acetate to Treat Wilson's Disease in Japan.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-02-2
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Wilson's Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NPC-02 (Experimental): zinc acetate
  Interventions: Drug: NPC-02

INTERVENTIONS:
Drug: NPC-02 — zinc acetate

SUMMARY:
The purpose of this long-term study is to determine whether Zinc Acetate is effective and safe in the treatment of Wilson's disease among Japanese.

DETAILED DESCRIPTION:
Wilson disease is an autosomal recessive disorder with copper metabolism. In Japan, the standard treatment is the use of copper chelating agents, such as D-penicillamine and trientine. In this study, we investigate efficacy on zinc acetate in Japanese patients with Wilson disease.

ELIGIBILITY:
Inclusion Criteria:

* Wilson's disease(adult, infant, pregnant woman)

Exclusion Criteria:

* Acute hepatitis
* Malignant tumor

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-03; Primary Completion 2008-04 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koudou Ishii, M.D., Study Director — National MINAMIYOKOHAMA Hospital

REFERENCES:
- [Result] Shimizu N, Fujiwara J, Ohnishi S, Sato M, Kodama H, Kohsaka T, Inui A, Fujisawa T, Tamai H, Ida S, Itoh S, Ito M, Horiike N, Harada M, Yoshino M, Aoki T. Effects of long-term zinc treatment in Japanese patients with Wilson disease: efficacy, stability, and copper metabolism. Transl Res. 2010 Dec;156(6):350-7. doi: 10.1016/j.trsl.2010.08.007. Epub 2010 Sep 23. PMID 21078496

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NPC-02
Started | 37
Completed | 34
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — A change of address | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed subjects comprised 37 patients who were found to have Wilson disease through clnical and biochemical tests.
Arm/Group | NPC-02
Number analyzed (Participants) | 37
Age, Customized [Number; unit: participants]
  ≥16 | 20
  ≥6 - <16 | 15
  ≥1 - <6 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Safety and Efficacy
Description: Number of patients who have at least one adverse events. ALT Change
Time Frame: During study period (up to 96W )
Population: The analysis was performed based on FAS population
Measure: Number; unit: participants
Arm/Group | NPC-02
Number analyzed (Participants) | 37
participants | 37

ADVERSE EVENTS:
Arm/Group | NPC-02
Serious Adverse Events (participants affected / at risk) | 4/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPC-02 (N=37)
Depression (Psychiatric disorders) | 1 (1)
Colitis ulcerative (Immune system disorders) | 1 (2)
Varicella (Infections and infestations) | 1 (1)
Sebaceous naevus (Congenital, familial and genetic disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPC-02 (N=37)
Conjunctivitis allergic (Eye disorders) | 2 (2)
Myopia (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 6 (6)
Stomach discomfort (Gastrointestinal disorders) | 7 (9)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Pain chest (General disorders) | 2 (2)
Edema peripheral (General disorders) | 2 (2)
Fever (General disorders) | 5 (5)
Seasonal allergy (Immune system disorders) | 2 (2)
Acute bronchitis (Infections and infestations) | 4 (5)
Gastroenteritis (Infections and infestations) | 4 (5)
Hordeolum (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 9 (9)
Molluscum contagious (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 24 (43)
Otitis meda (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 7 (7)
Rhinitis (Infections and infestations) | 3 (4)
Sinusitis (Infections and infestations) | 3 (3)
Varicella (Infections and infestations) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 2 (2)
Bruise (Injury, poisoning and procedural complications) | 2 (2)
ALT increased (Investigations) | 6 (6)
AST increased (Investigations) | 3 (3)
Blood alubumin decreased (Investigations) | 2 (2)
Blood amylase increased (Investigations) | 21 (23)
Blood bilirubin increased (Investigations) | 4 (4)
Cholesterol blood decreased (Investigations) | 6 (6)
Blood iron decreased (Investigations) | 22 (25)
Blood triglycerides increased (Investigations) | 12 (14)
Haematocrit decreased (Investigations) | 3 (3)
Blood urine present (Investigations) | 14 (15)
Hemoglobin decreased (Investigations) | 4 (4)
Lipase increased (Investigations) | 28 (29)
Mean cell haemoglobin concentration decreased (Investigations) | 4 (4)
Mean corpuscular volume decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 2 (3)
Protein total decreased (Investigations) | 2 (2)
White blood cell count decreased (Investigations) | 7 (7)
White blood cell count increased (Investigations) | 5 (5)
Platelet count increased (Investigations) | 3 (3)
Protein urine present (Investigations) | 13 (16)
Urobilin urine present (Investigations) | 2 (2)
ALP increased (Investigations) | 4 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 13 (19)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the sponsor and PI that no restricts the PI's right but need to discuss the timing of publish date of trial results after the trial is completed.